CLINICAL TRIAL: NCT04315727
Title: Identification of the Genetic Causes of Rare Diseases With Negative Exome Findings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GENOME +
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Rare Diseases; Genetic Predisposition to Disease
Keywords: Rare Diseases; Genetic Predisposition; Whole Exome Sequencing; Whole Genome Sequencing (WGS); WGS-trio analysis
MeSH Terms: conditions — Rare Diseases; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Other): Both underage and adult persons (male and female) with diagnostically unsolved rare diseases who have been or are included into diagnostic care at the University Hospital Tübingen, Germany (UKT) and who are suspected of having a genetic cause of the disease. In addition, healthy parents of volunteers will be recruited if available to facilitate Trio studies.
  Study related procedures: Blood sampling, hair collection, anamnesis including pedigree, Next Generation Sequencing (NGS) analysis and other omics analysis (transcriptomics, proteomics, metabolomics), functional cell biology studies (for example in fibroblast cultures, organoid cultivation).
  Interventions: Genetic: WGS Diagnostic Blood take for genetic diagnostic.; Genetic: Hair collection

INTERVENTIONS:
Genetic: WGS Diagnostic Blood take for genetic diagnostic. — Blood sampling, shot clinical characterization, WGS based trio sequencing, NGS analysis and other omics analysis (transcriptomics, proteomics, metabolomics), functional cell biology studies (for example in fibroblast cultures), RNA Sequencing (RNA-seq).
Genetic: Hair collection — Hair including root will be collected from the scalp (~15-20) and transferred to cultivation medium for the organoid cultivation

SUMMARY:
The GENOME + project will enroll patients (n = ca. 100) and their healthy parents with unclear molecular cause of the disease, suspected genetic cause of the disease and previous detailed molecular analysis like Whole Exome Sequencing (WES) did not lead to the identification of the disease causing mechanism. As well healthy parents of those affected for trio analysis (exception of one parent is not available for the study).

DETAILED DESCRIPTION:
In the GENOME+ study (monocentric, prospective, open-label diagnostic study), patients with molecularly undiagnosed diseases will diagnostically be analyzed by means of omics technologies or re-analyzed using existing datasets. The following questions will be leading the study:

Primary:

• Identification of the molecular causes of unclear rare diseases

Secondary:

* Improve number of diagnoses for patients with rare diseases
* Further characterization of the identified putative disease causes
* Increase number of patients receiving appropriate therapy after successful diagnosis.

In addition, healthy parents of the subjects may be included in the study to perform parent-child (trio) analyses.

In addition, phenotype and omics data will be shared within the University Hospital Tübingen, Germany and with external collaborators to improve the diagnostic rate of the patients included in the study.

Storage of blood or tissue samples is not primary goal of this project, but may be necessary for further analyses.

ELIGIBILITY:
Inclusion Criteria:

* Unclear diagnosis
* Suspected genetic cause of the disease
* Previous detailed molecular analysis like Whole Exome Sequencing (WES) did not lead to the identification of the disease causing mechanism
* Healthy parents of those affected for trio analysis (exception of one parent is not available for the study)

Exclusion Criteria:

* Missing informed consent of the patient and her/his parents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Identification of the molecular causes of unclear rare diseases | Day 1
  Number of molecular causes

SECONDARY OUTCOMES:
Diagnoses for patients with rare diseases | Day 1
  Number of diagnoses for patients with rare diseases
Molecular characterization of putative disease causes | Day 1
  Identify molecular characterization of the putative disease causes
Patients receiving appropriate therapy after successful diagnosis | Day 1
  Number of patients receiving appropriate therapy after successful diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Rieß, Study Director — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The GENOME+ study will provide data in a pseudonymized manner to national and international databases set up to increase the diagnostic yield through advanced analysis tools and matchmaking against other cohorts
Supporting Information: Analytic Code
Time Frame: Data will become available after analysis and unlimited.
Access Criteria: Authorized users within the participating organizations